CLINICAL TRIAL: NCT02707731
Title: Acute Effects of Neonatal Hydrokinesiotherapy in Newborn Preterm Hospitalized
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Pedro Ernesto (Other)
Responsible Party: Principal Investigator, Welcy Cassiano de Oliveira Tobinaga, Principal Investigator, Hospital Universitario Pedro Ernesto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUPedroernesto
Record Dates: First submitted 2016-03-03; First posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Newborn Preterm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydrokinesiotherapy in preterm (Experimental): Salivary cortisol samples, pain applying the Neonatal Infant Pain Scale Scale, heart rate, respiratory rate and oxygen saturation were collected before and after hydrokinesiotherapy
  Interventions: Procedure: Hydrokinesiotherapy

INTERVENTIONS:
Procedure: Hydrokinesiotherapy — physical therapy technique used in a plastic bucket approved by ANVISA , with water temperature monitored at 37 ° C, water level up to the shoulders and by the physical properties of water, was allowed to mobilize the newborn facilitating the feeling of relaxation and standard suitable movement.

SUMMARY:
This study aims to evaluate the acute effects of neonatal hydrokinesiotherapy in reducing stress in newborn preterm infants in the neonatal intensive care unit. Salivary cortisol samples were collected, pain applying the Neonatal Infant Pain Scale Scale (NIPS), heart rate, respiratory rate and oxygen saturation before and after hydrotherapy.

DETAILED DESCRIPTION:
Newborns have the neurological maturity to perceive pain, including preterm. In the environment of the neonatal intensive care unit newborns are subject to environmental stress and numerous painful interventions. Based on the physiological properties of water, it is known that the hydrotherapy promotes comfort, reduces stress, and as a resource for treatment of various diseases. This study aims to evaluate the acute effects of neonatal hydrokinesiotherapy in reducing stress in newborn preterm infants in the neonatal intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* gestational age above 37 weeks
* clinically stable
* without ventilatory support

Exclusion Criteria:

* access deep below the shoulders
* umbilical catheterization
* neurological and cardiac disorders
* clinically unstable

Max Age: 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Acute effects of heart rate after hydrokinesiotherapy in newborns preterm hospitalized | 4 months
  Unrecognized Condition
Acute effects of respiratory rate after hydrokinesiotherapy in newborns preterm hospitalized | 4 months
  Unrecognized Condition
Acute effects of salivary cortisol after hydrokinesiotherapy in newborns preterm hospitalized | 4 months
  Unrecognized Condition
Acute effects of peripheral oxygen saturation after hydrokinesiotherapy in newborns preterm hospitalized | 4 months
  Unrecognized Condition

SECONDARY OUTCOMES:
Acute effects of scale NIPS after hydrokinesiotherapy in newborns preterm hospitalized | 4 months
  Unrecognized Condition

CONTACTS AND LOCATIONS:
Overall Officials: Welcy Cassiano Tobinaga, Student, Principal Investigator — University Hospital Pedro Ernesto
Locations (1):
- Welcy Cassiano Tobinaga, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Oliveira Tobinaga WC, de Lima Marinho C, Abelenda VL, de Sa PM, Lopes AJ. Short-Term Effects of Hydrokinesiotherapy in Hospitalized Preterm Newborns. Rehabil Res Pract. 2016;2016:9285056. doi: 10.1155/2016/9285056. Epub 2016 Sep 8. PMID 27672453